CLINICAL TRIAL: NCT01662453
Title: Risk Factors for Sudden Unexplained Death in Epilepsy (SUDEP)
Brief Title: Risk Factors for Sudden Unexplained Death in Epilepsy
Acronym: SUDEP
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01664
Record Dates: First submitted 2012-08-02; First posted 2012-08-10 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: SUDEP
Keywords: epilepsy; seizures; mortality; sudep; risk factors
MeSH Terms: conditions — Sudden Unexpected Death in Epilepsy; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — If the family is willing to donate tissue, the family's permission is recorded in writing and it is filed in the subject's study record. The family can contact Autism Tissue Program (ATP) themselves or we will transfer the call to the ATP for them. The ATP has a 24/7 on call duty in place to receive new donors. The ATP coordinator will facilitate the donation process by coordinating with the family, medical examiner's office or hospital. The coordinator will also communicate to the research assistant when the donation is complete. In the case the participant does not want to donate tissue, but would like to donate other DNA samples, they will be able to do so through the NYU Biorepository. The participant will be consented, by research personnel, with the specific DNA collection consent form. Mucosal swaps or blood samples will be collected if available, if neither is available, we will collect hair or nails.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SUDEP Group: The SUDEP group refers to epileptic patients that had a sudden unexplained death; excludes trauma, drowning, status epilepticus, or other known cause, but there is often evidence of an associated seizure.
- Control Group: We will recruit living patients with epilepsy for the control group. In particular, epileptic patients with Dravet Syndrome of Idic 15.

SUMMARY:
The main purpose of this study is to develop a North American registry for SUDEP cases; requesting family members of epilepsy patients who died suddenly of unclear causes (SUDEP) to contact the study team. The family members who decide to participate in the study will be asked to complete a brief telephone interview about their loved one's epilepsy and seizure history and the circumstances of his or her death. If the death has occurred within the past 24 hours, and the family is willing to consider donating tissue to the study, the subject will be transferred to the Autism Tissue Program, and the remainder of the phone interview will be conducted at a later time.

In addition to the phone interview, the family will be asked to provide access to the deceased's medical records. Any costs involved in obtaining medical records will be covered by the study, and all medical information will remain completely confidential.

DETAILED DESCRIPTION:
SUDEP stands for sudden unexplained death in epilepsy; a witnessed or unwitnessed, non-traumatic and non-drowning death occurring in benign circumstances, in a person with epilepsy with or without evidence of a seizure and excluding documented status epileptics (seizure duration of 130mins or longer, or seizures without recovery in between), in which a postmortem examination does not reveal a cause of death. SUDEP is not a cause of death so much as it is a descriptive term for a category of unexplained deaths in people with epilepsy or epilepsy-related conditions. Little is known about SUDEP and its mechanisms and risk factors.

One of the main objectives of this study is to investigate the role of various risk factors in the development of sudden unexplained death in patients with epilepsy, with a particular focus on the role of antiepileptic medications. In addition, we want to elucidate the pathophysiologic mechanisms leading to SUDEP.

ELIGIBILITY:
Inclusion Criteria Sudep Group Subjects diagnosed with epilepsy whose cause of death was sudden and unexplained, and whose families are willing to participate, will be included in the study.

Control Group For the control group, we will include any patient diagnosed with epilepsy currently in the care of the NYU Comprehensive Epilepsy Center, willing and able to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The SUDEP group consists of epileptic patients who had a sudden unexplainable death excluding trauma, drowning, status epilepticus, or other known cause, but there is often evidence of an associated seizure.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-06; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
- Incidence of SUDEP - Risk factors for SUDEP. | 3 years
  Number of incidents of sudden unexplained deaths in epilepsy patients (SUDEP) and types of risk factors for SUDEP.

CONTACTS AND LOCATIONS:
Overall Officials: Orrin Devinsky, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Comprehensive Epilepsy Center, New York, New York, United States